CLINICAL TRIAL: NCT05249036
Title: Arterial Cannulation With Ultrasound
Acronym: ArCanUS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary event rate far higher than estimated for sample size calculation.
Sponsor: Queen Mary University of London (Other)
Collaborators: The London Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 301584
Record Dates: First submitted 2022-01-26; First posted 2022-02-21 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Perioperative/Postoperative Complications
Keywords: Arterial cannulation; Ultrasound
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guided arterial cannulation (Experimental): Anaesthetist will use real-time ultrasound guidance to guide arterial cannulation
  Interventions: Procedure: Ultrasound guided arterial cannulation
- Palpation guided arterial cannulation (Active Comparator): Anaesthetist will use palpation (standard-of-care) technique to guide arterial cannulation
  Interventions: Procedure: Palpation guided arterial cannulation

INTERVENTIONS:
Procedure: Ultrasound guided arterial cannulation — Arterial cannulation will be attempted at the site of the radial artery of the non-dominant hand, using real-time ultrasound guidance
  Arms: Ultrasound guided arterial cannulation
Procedure: Palpation guided arterial cannulation — Arterial cannulation will be attempted at the site of the radial artery of the non-dominant hand, using palpation technique (standard-of-care)
  Arms: Palpation guided arterial cannulation

SUMMARY:
A drop in blood pressure during anaesthesia for a surgical procedure has been associated with worse patient outcomes, including complications such as damage to the heart, brain and kidneys. Continuous blood pressure monitoring prior to the start of anaesthesia alerts the anaesthetist to drops in blood pressure and allows this to be treated promptly. This may help to avoid the complications described above.

Continuous blood pressure monitoring is carried out by inserting a small plastic tube (cannula) into an artery. In this study, the investigators propose inserting a cannula into the radial artery in the wrist before a patient is anaesthetised for surgery. The usual technique for insertion of this cannula is for the anaesthetist to identify the site of the radial artery by feeling for an arterial pulse with the fingertips (palpation). An alternative technique for identification is to use ultrasound. Ultrasound creates a two-dimensional image of the area under the skin on a screen, enabling the operator to visualise the artery being targeted. This may reduce the number of cannulation attempts required, reducing patient discomfort.

DETAILED DESCRIPTION:
The investigators will test whether ultrasound guidance improves the success rate of radial artery cannulation, compared to palpation alone, in a randomised controlled trial in an NHS hospital. Patients will be over 45 years old, undergoing general or neuraxial anaesthesia for non-cardiac surgery lasting 120 minutes or more. Patients will be randomly assigned to a palpation or ultrasound-guided technique for arterial cannulation. Patients will receive numbing local anaesthetic cream to the area beforehand. A needle is used to introduce the cannula into the artery. There will be a maximum of one attempt allowed. In addition to measuring success rate, we will also compare whether the successfully sited cannula provides an adequate arterial waveform, requires resiting at any point during the surgery and any complications which arise directly related to arterial catheterisation. Patients will receive standard anaesthetic and surgical care in all other respects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled to undergo major elective or urgent (not requiring intervention in <24 hours) non-cardiac surgery under general anaesthesia and/or neuraxial anaesthesia, expected to take >120 minutes from induction of anaesthesia
2. Requiring overnight hospital stay.

Exclusion Criteria:

1. Anatomical deformity
2. Unable to consent
3. Cannulation attempt within 24 hours
4. Overlying infection

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-12-25 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Success rate at first attempt to cannulate the radial artery | 10 minutes
  Success is defined as radial artery cannulation resulting in a transduced arterial waveform. First attempt is defined as one needle puncture through the skin.

SECONDARY OUTCOMES:
Characteristics of arterial waveform | Within 15 mins of catheterisation.
  Assessment for presence of: (1) Dicrotic notch; (2) >1 oscillation after fast flush; (3) <3 oscillations after fast flush
Complications | 24 hours
  Recannulation required before/after surgery, infection, hematoma, thrombus.

CONTACTS AND LOCATIONS:
Overall Officials: Gareth L Ackland, PhD FRCA, Principal Investigator — Translational Medicine & Therapeutics, William Harvey Research Institute, Barts and The London School of Medicine and Dentistry, Queen Mary University of London
Locations (1):
- Royal London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lan-Pak-Kee V, Ackland GL, Egan TC, Abbott TE, Elsheikh F; Arterial Cannulation with Ultrasound Investigators. Arterial cannulation with ultrasound: clinical trial protocol for a randomised controlled trial comparing handheld ultrasound versus palpation technique for radial artery cannulation. BJA Open. 2022 Dec;4:None. doi: 10.1016/j.bjao.2022.100111. PMID 36561483